CLINICAL TRIAL: NCT01023503
Title: Statins Use Patterns in Spain
Brief Title: Observational Study To Evaluate Statins Patterns Of Use In Spain
Status: Withdrawn | Type: Observational
Why Stopped: Changes affecting Post Authorization Study Regulatory effective from Dec09, impacted the requirements for Spanish studies at National and Regional level.
Sponsor: AstraZeneca (Industry)
Collaborators: Fundació Institut Català de Farmacologia (Unknown)
Responsible Party: Sponsor
Other Study IDs: NIS-CES-CRE-2009/1
Record Dates: First submitted 2009-10-31; First posted 2009-12-02 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Dyslipidemia
Keywords: Statins; Dyslipidemia; Spain; Rosuvastatin; Naive; Switching; New statins prescriptions in Spain (naive patients and switching)
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Adults, with a new statin prescription or a change in their stain treatment

SUMMARY:
The present project is aimed at describing the statins prescription pattern in Spanish patients. It will also look into how adequate these prescriptions are accordingly to the recommendations given in Treatment Guidelines and in the Summary Product Information.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving a new statin prescription (naïve patients)
* Patients having a change in their statin prescription (dose, switching, addition to another hypolipemic drug)

Exclusion Criteria:

* Patients without enough information in the medical records to complete the fields required in the eCRF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To be recruited by Primary Care Physicians
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2012-04 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Current and previous hypolipemic treatment, dose and pattern | Retrospectively (information for the previous 6-months). Information collected once.
Statin treatment start date, origin of the prescription, reasons for changes in prescription | Retrospectively (information for the previous 6-months). Information collected once.

SECONDARY OUTCOMES:
Socio-demographic characteristics | retrospectively
Total Cholesterol, HDL, LDL, Triglycerides, ALAT, Glucose, Creatine Kinase plasma levels | retrospectively
Concomitant Treatments and Cardiovascular History | retrospectively

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Barcelona, Spain